CLINICAL TRIAL: NCT05994898
Title: The Value of Ultrahigh-frequency Ultrasonography (UHFUS) in Detection of Small Pulmonary Ground Glass Opacity (GGO) in Vitro: A Prospective Pilot Study
Brief Title: Ultrahigh-frequency Ultrasonography (UHFUS) in Detection of Small Pulmonary Ground Glass Opacity (GGO)
Acronym: UHFUSGGO
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xuehan Gao, MD, Peking Union Medical College Hospital
Other Study IDs: UHFUSGGO01
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lung Nodules; Ultrasound; Detection Rate
Keywords: lung nodules; ground glass opacity; Ultrahigh frequency ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UHFUS: Pulmonary nodules were detected by UHFUS method.
- Palpation: Pulmonary nodules were detected by palpation method.

SUMMARY:
The purpose of this study is to assess the feasibility of UHFUS on detection of GGOs in excised lung tissue and investigate UHFUS features of GGO in vitro.

Each GGO was detected by palpation, UHFUS and open biopsy in sequence. The comparison of detection rate and time consumption were analyzed respectively. The Bland-Altman analysis was used to estimate the agreement of tumor size measured by CT, UHFUS and pathology.

DETAILED DESCRIPTION:
Lung cancer (LC) is a leading cause of mortality worldwide. According to the International Agency for Research (IARC) on Cancer, LC was projected to contribute to 2.3 million new cancer cases and 1.8 million deaths worldwide in 2020. With widespread use of chest computed tomography (CT), LC is increasingly detected at an early stage, in which 63%-95% lesions present as ground glass opacity (GGO).

GGO refers to a non-specific radiological appearance, referring to a focal, hazy shadow with increased attenuation that does not obscure the contours of bronchi or blood vessels on CT. It can be benign lesions, preinvasive, or invasive adenocarcinoma. Surgery is the main treatment for suspected malignant GGOs. Whether excised targeted GGOs thoroughly affects patients' prognosis crucially, especially for patients with multiple GGOs. Generally, the most frequent intraoperative location approach of pulmonary nodules is palpation, which distinguished by the texture between normal lung tissue and nodules. However, different from solid nodules, the texture of GGO nodules is similar to lung parenchyma that increases the difficulty of palpation localization. Thus, detection of GGOs and in lung tissue poses a common challenge, particularly in the presence of pure GGO (tumor without an solid component) and small GGO nodules (≤1cm).

In the current clinical practice, even with preoperative localization (CT-guided percutaneous and intraoperative electromagnetic navigation bronchoscopy), it remains challenging to confirm complete resection of all small, pure GGOs. Therefore, there is an urgent need for a new method that can accurately evaluate nodules in excised lung tissue. Since Roberto used thoracoscopic ultrasound (TUS) to examine pulmonary nodules in 1999, subsequently, several studies have validated the safety and efficacy for using US in identifying pulmonary nodules intraoperatively. However, past research all focused on solid nodules or large nodules (maximum diameter more than 2cm) using 5-12MHz US transducer. Few studies have studied the detection rate of small GGO nodules.

Previous studies have found 12MHz of US probe could show pulmonary nodules better than 5MHz and 7.5MHz. Ultrahigh frequency ultrasound (UHFUS) refers to higher frequency (≥20MHz) ultrasound waves with higher resolution even less than 50μm. It is capable to display nodules less than 3mm distinctively in the extremely superficial tissue, which may satisfy intraoperative GGO imaging requirement. Therefore, the objects of this study are to assess the feasibility of localizing GGOs in excised lung tissue by UHFUS and further summarize its UHFUS features.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with targeted nodules identified as lesions required surgical removed such as main lesion and high-risk nodules;
2. Patients who accept VATS or RATS resection.

Exclusion Criteria:

1. Patients refused enrollment in the trial;
2. Pulmonary nodules were labelled during the operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with targeted GGOs and will accept VATS or RATS resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection rate | From enrollment to the pathology of GGOs were confirmed (4 weeks after sugery)
  Detection rate of UHFUS and palpation methods

SECONDARY OUTCOMES:
Detection time | From enrollment to the end of surgery
  Detection time of UHFUS and palpation methods

OTHER OUTCOMES:
UHFUS imaging features | From enrollment to the end of surgery
  UHFUS imaging features of GGOs
Tumor size | From enrollment to the pathology of GGOs were confirmed (4 weeks after sugery)
  The agreement of tumor size measured by CT, UHFUS and pathology

CONTACTS AND LOCATIONS:
Overall Officials: Shanqing Li, Prof., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of thoracic surgery, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, SAP, and ICF could be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after the trial finnshed.
Access Criteria: Contact investigators by email (GXH: gaoxh1299@163.com, GYJ: 610066214@qq.com).

REFERENCES:
- [Background] Ujiie H, Kato T, Hu HP, Hasan S, Patel P, Wada H, Lee D, Fujino K, Hwang DM, Cypel M, de Perrot M, Pierre A, Darling G, Waddell TK, Keshavjee S, Yasufuku K. Evaluation of a New Ultrasound Thoracoscope for Localization of Lung Nodules in Ex Vivo Human Lungs. Ann Thorac Surg. 2017 Mar;103(3):926-934. doi: 10.1016/j.athoracsur.2016.08.031. Epub 2016 Oct 17. PMID 27765176
- [Background] Yamamoto M, Takeo M, Meguro F, Ishikawa T. Sonographic evaluation for peripheral pulmonary nodules during video-assisted thoracoscopic surgery. Surg Endosc. 2003 May;17(5):825-7. doi: 10.1007/s00464-002-8900-0. Epub 2003 Jan 18. PMID 12584601
- [Background] Sortini D, Feo CV, Carcoforo P, Carrella G, Pozza E, Liboni A, Sortini A. Thoracoscopic localization techniques for patients with solitary pulmonary nodule and history of malignancy. Ann Thorac Surg. 2005 Jan;79(1):258-62; discussion 262. doi: 10.1016/j.athoracsur.2004.06.012. PMID 15620953
- [Background] Wada H, Anayama T, Hirohashi K, Nakajima T, Kato T, Waddell TK, Keshavjee S, Yoshino I, Yasufuku K. Thoracoscopic ultrasonography for localization of subcentimetre lung nodules. Eur J Cardiothorac Surg. 2016 Feb;49(2):690-7. doi: 10.1093/ejcts/ezv124. Epub 2015 Apr 7. PMID 25855597
- [Background] Santambrogio R, Montorsi M, Bianchi P, Mantovani A, Ghelma F, Mezzetti M. Intraoperative ultrasound during thoracoscopic procedures for solitary pulmonary nodules. Ann Thorac Surg. 1999 Jul;68(1):218-22. doi: 10.1016/s0003-4975(99)00459-2. PMID 10421144
- [Background] Matsunaga T, Suzuki K, Takamochi K, Oh S. What is the radiological definition of part-solid tumour in lung cancer?dagger. Eur J Cardiothorac Surg. 2017 Feb 1;51(2):242-247. doi: 10.1093/ejcts/ezw344. PMID 28119328
- [Background] Hou YL, Wang YD, Guo HQ, Zhang Y, Guo Y, Han H. Ultrasound location of pulmonary nodules in video-assisted thoracoscopic surgery for precise sublobectomy. Thorac Cancer. 2020 May;11(5):1354-1360. doi: 10.1111/1759-7714.13384. Epub 2020 Mar 17. PMID 32180358
- [Background] Zhang Y, Fu F, Chen H. Management of Ground-Glass Opacities in the Lung Cancer Spectrum. Ann Thorac Surg. 2020 Dec;110(6):1796-1804. doi: 10.1016/j.athoracsur.2020.04.094. Epub 2020 Jun 7. PMID 32525031
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338